CLINICAL TRIAL: NCT00782288
Title: Phase II Study of Digitoxin to Treat Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Pam Zeitlin, Professor of Pediatrics, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FD-R-003456-01
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
Keywords: digitoxin; inflammatory markers; cytokines; gene expression
MeSH Terms: conditions — Cystic Fibrosis | interventions — Digitoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): low dose 0.05mg digitoxin given once daily for 28 days
  Interventions: Drug: digitoxin
- 2 (Active Comparator): higher dose 0.1mg digitoxin daily for 28 days
  Interventions: Drug: digitoxin
- 3 (Placebo Comparator): placebo given daily for 28 days
  Interventions: Other: placebo

INTERVENTIONS:
Drug: digitoxin — 0.05mg tabs, once daily for 28 days
  Arms: 1
Drug: digitoxin — 0.1mg pills, once daily for 28 days.
  Arms: 2
Other: placebo — pill taken once daily for 28 days
  Arms: 3

SUMMARY:
This study will measure the inflammatory effects of digitoxin on IL-8 and neutrophil counts in induced sputum in stable Cystic Fibrosis (CF) patients and the pharmacokinetics of digitoxin in serum.

Funding Source-FDA OOPD

DETAILED DESCRIPTION:
The study will be conducted as a randomized, double blind, placebo-controlled, repeat dosing trial evaluating the effects of 28 days of digitoxin on IL-8 and neutrophil concentrations in induced sputum in subjects with mild to moderate cystic fibrosis lung disease. Twenty-four total patients will be randomized into 3 groups of 8 subjects each (0.05 mg or 0.1 mg digitoxin or a placebo).

ELIGIBILITY:
Inclusion Criteria

* Male or female 18-45 years of age
* Confirmed diagnosis of CF based on the following criteria:positive sweat chloride > or = 60 mEq/liter (by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF
* FEV1 > or = 40% predicted value at screening
* Weight > 45 kg at Screening and Visit 1 (dosing)
* Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation (see Appendix II) or treatment of a pulmonary exacerbation within the 14 days prior to Screen Visit. Subject may rescreen 14 days after they complete treatment for a pulmonary exacerbation, if healthy at that time.
* Ability to perform Spirometry.
* Ability to understand and sign a written informed consent and comply with the requirements of the study.

Exclusion Criteria:

* Use of an investigational agent within the 4-week period prior to Screen visit.
* Use of a medication with anti-neutrophil or anti-inflammatory effect or those known to have an effect on inflammatory outcomes [azithromycin, gentamicin, amikacin, colistin, ibuprofen, celecoxib, or other NSAIDs, prednisone or other corticosteroids(systemic or inhaled), such as Advair, cromolyn (Intal®), montelukast (Singulair®), zafirlukast (Accolate®), zileuton (Zyflo®), and any immunosuppressive agent within the 4 weeks prior to Visit #1, Day 1 and until their participation in the study ends (after Visit 6). See NOTE at end of exclusionary criteria for subjects on oral antibiotic therapy.
* Use of topical nasal steroid products for at least 2 weeks prior to study drug administration and discontinued use until after the nasal cell collection at Day 28.
* Inability or unwillingness to stop macrolide antibiotics 4 weeks prior to Day 1 until their participation in the study ends. Prior use of macrolide antibiotics, including those for maintenance therapy will not exclude the subject from participation.
* History of significant cardiac disease or cardiac arrhythmia
* Presence of an arrhythmia identified on screening ECG or 24 hour holter monitor
* Pulmonary hypertension
* History of significant cardiac disease or cardiac arrhythmia
* Presence of a clinically significant arrhythmia identified on screening ECG or 24 hour holter monitor.
* Pulmonary hypertension
* Burkholderia species in sputum within 2 years or at Screen visit
* Drugs known to interact with digitoxin including phenobarbital, amphotericin B, rifampicin, diltiazem, and verapamil or drugs that would potentiate potassium loss (certain diuretics or excessive laxative use, defined as more than twice daily use of miralax).
* Unwillingness to use beta-agonists (or levalbuterol) prior to induced sputum procedures.
* Oxygen saturation < 92% on room air at Screen visit
* Pregnant, breastfeeding, or unwilling to use an effective form of birth control for the duration of the study
* History of significant hemoptysis > or = 60cc per episode during the 30 days prior to Screening visit
* Significant history of hepatic, cardiovascular, renal, neurological, hematologic, or peptic ulcer disease
* SGOT (ALT) or SGPT (AST) > 3 times the upper limit of normal at Screen, documented biliary cirrhosis, or portal hypertension
* Creatinine > 1.8 mg/dL at Screen
* Inability to swallow pills
* Potassium, serum <3.3 mEq/L at screening
* Known inability to produce sputum (if unable to expectorate, must be able to produce an induced sputum sample at screening).
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data NOTE: For subjects on continuous antibiotic therapy for at least 6 months one continuous antibiotic or alternating two different antibiotics, they can maintain their current therapy. If the subject is alternating between two different inhaled antibiotics each month, Visit 1 should coincide with the "on" cycle of one of the inhaled antibiotics for consistency during the treatment period. For subjects on alternate month TOBI®, colistin or Cayston therapy, the "off" cycle must coincide with the Treatment Phase of the study. Subjects should be scheduled for Screening Visit during their one-month "on" period, and may resume taking TOBI®, colistin or Cayston after completion of Visit 6 (Day 42) or early termination.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Zeitlin, MD, PhD, Principal Investigator — Johns Hopkins University, School of Medicine, Pediatric Pulmonary
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Zeitlin PL, Diener-West M, Callahan KA, Lee S, Talbot CC Jr, Pollard B, Boyle MP, Lechtzin N. Digitoxin for Airway Inflammation in Cystic Fibrosis: Preliminary Assessment of Safety, Pharmacokinetics, and Dose Finding. Ann Am Thorac Soc. 2017 Feb;14(2):220-229. doi: 10.1513/AnnalsATS.201608-649OC. PMID 28006108
- See also: Johns Hopkins Cystic Fibrosis website — http://www.hopkinscf.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the Johns Hopkins University in Baltimore, Maryland. The first participant was enrolled on October 13, 2010 and the last participant was enrolled on May 6, 2014. All study visits were completed as of June 2014. There was a DSMB safety review prior to enrolling any subjects into the higher dose group (0.1 mg).
Pre-assignment Details: Participants were all consented on a Johns Hopkins IRB approved consent form and screened 2 or 4 weeks prior to enrollment. Enrollment was contingent on meeting all inclusion/exclusion criteria.
Groups:
- Placebo: placebo given daily for 28 days
  placebo: pill taken once daily for 28 days
- Low Dose 0.05mg Digitoxin: low dose 0.05mg digitoxin given once daily for 28 days
  digitoxin: 0.05mg tabs, once daily for 28 days
- Higher Dose 0.1mg Digitoxin: higher dose 0.1mg digitoxin daily for 28 days
  digitoxin: 0.1mg pills, once daily for 28 days.
Period: Overall Study
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose 0.05 mg Digitoxin: low dose 0.05mg digitoxin given once daily for 28 days
  digitoxin: 0.05mg tabs, once daily for 28 days
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose 0.05 mg Digitoxin | Higher Dose 0.1mg Digitoxin | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.8 [18.2 to 39.7] | 23.5 [18.2 to 37.7] | 30.3 [19.8 to 42.8] | 26.2 [18.2 to 42.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 13
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Effect of Digitoxin on IL-8 (Interleukin 8) in Induced Sputum in Stable Cystic Fibrosis (CF) Patients.
Description: The Il-8 measurements of sputum digitoxin levels for each group is shown for 5 days (Days 1, 14, 21, 28 and 42).
Time Frame: 42 days (Day 1 to Day 42)
Population: Sputum was collected for Il-8 biomarkers on Days 1,14, 21, 28 during the treatment phase and at Day 42. Measures were compared between Baseline, Treatment and Recovery periods to determine if changes from baseline differed between placebo and the two doses.
Measure: Median (Inter-Quartile Range); unit: log 10 (pg/mL)
Arm/Group | Placebo | Low Dose 0.05 mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
log 10 (pg/mL)
  IL-8 Day 1 | 4.59 [4.15 to 5.12] | 4.96 [4.4 to 5.18] | 5.04 [4.58 to 5.10]
  IL-8 Day 14 | 4.94 [4.21 to 5.34] | 4.89 [4.50 to 5.01] | 5.01 [4.66 to 5.45]
  IL-8 Day 21 | 5.08 [4.21 to 5.38] | 4.77 [4.64 to 4.89] | 5.17 [4.66 to 5.42]
  IL-8 Day 28 | 4.66 [4.49 to 5.38] | 4.79 [4.49 to 4.91] | 5.20 [4.68 to 5.34]
  IL-8 Day 42 | 4.59 [4.22 to 5.06] | 4.74 [4.62 to 5.04] | 4.97 [4.43 to 5.25]
Statistical Analysis 1: Comparison: Placebo vs Low Dose 0.05 mg Digitoxin vs Higher Dose 0.1mg Digitoxin; Measures were compared between Baseline, Treatment & Recovery periods to determine if changes from baseline differed between placebo and the two digitoxin dose levels. Kruskal-Wallis equity of population rank test was performed on the changes Day 28 minus Day 1. To compare the change from baseline to treatment period between the two arms, a Wilcoxon rank sum test was performed. To determine whether induced sputum Il-8 returned to baseline at the final visit, a one sample sign test was performed; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pharmacokinetics (PK) of Digitoxin in Serum in Stable CF Patients.
Description: Digitoxin serum levels were drawn on Days 1 (pre-dose), 7, 14, 21 and 42. The range of digitoxin levels for each visit is listed and the number of subjects who had that level are marked by group (placebo, low dose and high dose).
Time Frame: Serum PK on Days 1 (pre-dose), 7, 14, 21 and 42
Population: Subjects had serum digitoxin levels drawn at Day 1 (pre-dose) with no levels observed, as expected. Digitoxin was drawn on Day 7, 14, 21 and 42 to determine the number of subjects with a detectable level of digitoxin (ng/mL) in serum by group.
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
participants
  Day 7, digitoxin level 5.6 ng/mL | 0 | 0 | 1
  Day 7, digitoxin level 6 ng/mL | 0 | 1 | 1
  Day 7, digitoxin level 6.4 ng/mL | 0 | 0 | 1
  Day 7, digitoxin level 6.9 ng/mL | 0 | 0 | 1
  Day 7, digitoxin level 7.8 ng/mL | 0 | 0 | 1
  Day 7, digitoxin level none detected | 8 | 7 | 3
  Day 14, digitoxin level 10 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 11 ng/mL | 0 | 1 | 0
  Day 14, digitoxin level 13 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 6.8 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 6.9 ng/mL | 0 | 1 | 0
  Day 14, digitoxin level 7.3 ng/mL | 0 | 1 | 0
  Day 14, digitoxin level 7.5 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 8.1 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 9.3 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level 9.4 ng/mL | 0 | 0 | 1
  Day 14, digitoxin level none detected | 8 | 5 | 1
  Day 21, digitoxin level 10 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 11 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 12 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 13 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 14 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 15 ng/mL | 0 | 1 | 0
  Day 21, digitoxin level 4 ng/mL | 0 | 1 | 0
  Day 21, digitoxin level 5 ng/mL | 0 | 1 | 0
  Day 21, digitoxin level 6 ng/mL | 0 | 1 | 0
  Day 21, digitoxin level 6.4 ng/mL | 0 | 1 | 0
  Day 21, digitoxin level 6.5 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 6.9 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level 7.5 ng/mL | 0 | 0 | 1
  Day 21, digitoxin level none detected | 8 | 3 | 0
  Day 42, digitoxin level 5 ng/mL | 0 | 1 | 0
  Day 42, digitoxin level none detected | 8 | 7 | 8

3. Secondary Outcome: Safety Indices Including Change in FEV1 in Stable CF Patients.
Description: Safety indices included changes in FEV1 (forced expiratory volume in 1 second), changes in WBC (white blood cell count), alterations in ECG and sputum microbiology. The median changes in FEV1 are reported.
Time Frame: Baseline and Day 28
Population: Median changes in FEV1 in L by group for the 28 days of treatment.
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
liters | -0.00 [-0.37 to 0.22] | 0.10 [0.05 to 0.13] | -0.02 [-0.14 to 0.07]

4. Secondary Outcome: Mean Change in Quality of Life Scores, for Each Domain, From Day 1 to Day 42 Using the Cystic Fibrosis Questionnaire Revised (CFQ-R).
Description: CFQ-R is a disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms. Developed specifically for use in patients with a diagnosis of cystic fibrosis. There are 9 Quality of life domains: physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions and 3 symptom scales: weight, respiratory, and digestion.
  Scaling of items is done via 5 distinct 4-point Likert scales. Scores for each domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health. Based on clinician judgment of global clinical change, a moderate change was a standardized effect size of 0.50 units and an important change was a standardized effect size of 0.80 units evaluating pre- and post-treatment for CF exacerbation. Mean changes in CFQ-R Scores by Group were evaluated between Visit 6 and Visit 1, by Domain.
Time Frame: Baseline and Day 42
Population: Mean change in CFQ-R scores from Visit 1 to Visit 6, by domain.
Measure: Mean (Standard Deviation); unit: mean change of scores on a scale
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
mean change of scores on a scale
  Physical Domain | -5.21 (8.55) | -14.58 (17.11) | -2.60 (11.34)
  Role Domain | 0.00 (7.72) | -1.04 (5.34) | 1.04 (8.26)
  Vitality Domain | -2.08 (5.89) | 4.17 (6.30) | 1.04 (20.62)
  Emotional Domain | -5.83 (12.57) | -5.00 (17.73) | 4.17 (13.30)
  Social Domain | -2.08 (9.36) | -5.56 (6.64) | -4.17 (15.92)
  Body Domain | 6.94 (14.47) | -4.17 (22.17) | 8.33 (11.50)
  Eating Domain | -1.39 (11.01) | -1.39 (3.93) | -1.39 (3.93)
  Treatment Domain | 1.39 (9.27) | 6.94 (11.79) | 5.56 (8.40)
  Health Domain | 1.39 (9.27) | 4.17 (5.75) | -4.17 (11.79)
  Weight Domain | 0.00 (0.00) | 12.50 (17.25) | -0.00 (17.82)
  Respiratory Domain | -2.78 (13.61) | 2.78 (13.28) | -6.94 (22.17)
  Digestion Domain | -9.72 (12.51) | 4.17 (10.18) | -5.56 (16.80)

5. Secondary Outcome: Change in WBC (White Blood Cell) Count by Group During Treatment Period
Description: Safety indices included changes in FEV1 (lung function), changes in WBC, alterations in ECG and sputum microbiology. There were no significant alterations in the ECG in any subjects over the course of the study. There were no subjects who acquired multiple resistant changes in microbiology of sputum and no acquisition of B. cepacia in any subjects. Therefore, these data were not analyzed. The median changes in FEV1 and median changes in WBC, ESR and CRP are reported.
Time Frame: Baseline and Day 28
Population: Safety indices included changes in WBC during treatment for each group.
Measure: Median (Inter-Quartile Range); unit: K/cu mm
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
K/cu mm | -510.28 [-2775.00 to 350.92] | -0.98 [-680.00 to 930.00] | -0.13 [-2130.63 to 1.87]

6. Primary Outcome: Change in Il-8 (Interleukin 8) Levels From Day 28 Minus Day 1 (Treatment Period).
Description: Change in Il-8 values are expressed as a change in log 10 Il-8 pg/mL from Day 28 minus Day 1.
Time Frame: 28 days (Day 28 minus Day 1)
Population: For change in Il-8 from Day 28 minus Day 1, a Kruskal-Wallis equality of populations rank was performed.
Measure: Median (Inter-Quartile Range); unit: log10 (pg/mL)
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
log10 (pg/mL) | 0.13 [0.06 to 0.40] | -0.13 [-0.23 to 0.16] | 0.04 [-0.24 to 0.41]

7. Primary Outcome: Effect of Digitoxin on Neutrophil Counts in Induced Sputum in Stable Cystic Fibrosis (CF) Patients.
Description: The neutrophil counts were measured in the induced sputum of participants in each group on study 5 days (Days 1, 14, 21, 28 and 42).
Time Frame: 42 days (Day 1- Day 42)
Population: Neutrophil cell counts were compared between Baseline, Treatment and Recovery periods to determine if changes from baseline differed between the placebo and the two digitoxin dose levels.
Measure: Median (Inter-Quartile Range); unit: log 10 (neutrophil cells/mL)
Arm/Group | Placebo | Low Dose 0.05 mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 7 | 7
log 10 (neutrophil cells/mL)
  Day 1 | 2.58 [1.89 to 3.00] | 2.82 [1.88 to 3.08] | 2.93 [2.35 to 3.04]
  Day 14 | 2.89 [2.18 to 2.92] | 2.26 [1.35 to 2.91] | 2.71 [2.26 to 3.10]
  Day 21 | 2.86 [2.44 to 3.35] | 2.23 [1.52 to 2.62] | 2.88 [1.90 to 3.14]
  Day 28 | 2.71 [2.16 to 3.06] | 2.16 [0.83 to 2.64] | 2.77 [1.97 to 3.01]
  Day 42 | 2.55 [2.27 to 2.81] | 2.06 [1.58 to 2.35] | 2.82 [2.00 to 2.96]
Statistical Analysis 1: Comparison: Placebo vs Low Dose 0.05 mg Digitoxin vs Higher Dose 0.1mg Digitoxin; Baseline,Treatment and Recovery periods were compared to determine if changes from baseline differed between placebo and the two digitoxin doses; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Change in Neutrophil Cell Count Day 28 Minus Day 1 (Treatment Period).
Description: The change in log 10 neutrophil cell count from Day 28 minus Day 1 (during the treatment period) expressed as log (10^4 neutrophil/mL).
Time Frame: 28 days (Day 28 minus Day 1)
Population: The change in neutrophil cell count from Day 1 to Day 28 was performed using a Kruskal-Wallis equality of populations rank test. The cells counts are expressed as log 10 (neutrophil cell/mL).
Measure: Median (Inter-Quartile Range); unit: log 10 (neutrophil cell/mL)
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 7 | 7
log 10 (neutrophil cell/mL) | 0.19 [-0.24 to 0.82] | -0.26 [-0.41 to 0.29] | -0.02 [-0.33 to 0.26]

9. Secondary Outcome: Changes in C Reactive Protein (CRP) During Treatment.
Description: Median changes in CRP and IQR were assessed from serum samples collected at Visits 1,3, 4 and 5.
Time Frame: Baseline and Day 28
Population: All subjects had blood labs for CRP drawn on Visits 1,3,4 and 5. The changes in median CRP were calculated during the Treatment Period (28 days).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
mg/dL | -0.20 [-0.50 to 0.15] | 0.05 [0.00 to 0.40] | -0.05 [-0.20 to 0.05]

10. Secondary Outcome: Changes in Erythrocyte Sedimentation Rate (ESR) During Treatment Period.
Description: Median change in serum ESR (mm/hr) and IQR was calculated from Treatment Period (28 days).
Time Frame: Baseline and Day 28
Population: All subjects had blood labs for ESR drawn on Visits 1,3,4 and 5. The changes in median ESR were calculated during the Treatment Period (28 days).
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
mm/hr | -1.00 [-5.50 to 0.50] | 3.50 [0.05 to 11.50] | 0.00 [-3.50 to 5.00]

11. Secondary Outcome: Number of CF Subjects With Microarray Results From Nasal Epithelial Cells to Measure the Effect of Digitoxin on Gene Expression.
Description: Rhinoprobe was used to collect nasal epithelial cells. The cells were collected pre and post-treatment and placed in Trizol for RNA isolation then used to measure the effect of digitoxin on gene expression. The full set of microarray data has been deposited in the National Center for Biotechnology Information (NCBI) Gene Expression Omnibus (GEO). The accession number for that data is GSE76347 (data available Dec 2018).
Time Frame: Day 0 and Day 28
Population: The full set of microarray data has been deposited in the National Center for Biotechnology Information (NCBI) Gene Expression Omnibus (GEO). Results can be found under the accession number GSE76347. One subject's pair of specimens in the placebo group was not collected.
Measure: Number; unit: participants
Groups:
- All Participants: All study participants had nasal cells collected pre and post treatment during the study. Because the data set is extremely large, the full set of microarray data has been deposited in the National Center for Biotechnology Information (NCBI) Gene Expression Omnibus (GEO) this information can be obtained under the accession number.
Arm/Group | All Participants
Number analyzed (Participants) | 23
participants | 23

12. Secondary Outcome: Clinically Significant Alterations in ECG Readings
Description: Safety indices included an assessment for the number of clinically significant alterations in the subjects ECG readings from Day 1 to Day 28.
Time Frame: 28 days
Population: Count of clinically significant alterations in the ECG in all subjects during the Treatment Phase of the study.
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

13. Secondary Outcome: Clinically Significant Changes in the Microbiology of Sputum in Subjects
Description: Count of clinically significant changes in sputum microbiology during the Treatment phase (Day 1 to Day 28) to include any new acquisition of B. cepacia or new acquisition of any multiple resistant organism.
Time Frame: 28 days
Population: There were no significant changes in the microbiology of sputum in any subjects over the course of treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose 0.05mg Digitoxin | Higher Dose 0.1mg Digitoxin
Number analyzed (Participants) | 8 | 8 | 8
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Screening through Day 42 or the Early Withdraw Visit.
Description: Physical exams by study physician at each visit and documented in the subject case report forms. All Adverse Events were subsequently followed up until resolution.
Arm/Group | Placebo | Low Dose 0.05 mg Digitoxin | Higher Dose 0.1mg Digitoxin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 5/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Low Dose 0.05 mg Digitoxin (N=8) | Higher Dose 0.1mg Digitoxin (N=8)
abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1)
anxiety (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
chills (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
decrease breath sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
decreased lung function (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
epistaxis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
erythema, nares (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1) | 1 (2)
fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
headache (General disorders) | 3 (3) | 4 (8) | 3 (3)
hemoptysis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
increased sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
increased urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1)
pain, nares (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
night sweats (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
sore throat (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
tonic clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
wheeze (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
vaginal yeast infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Steady states of digitoxin were not achieved in subjects until relatively late the in 28 day treatment period. This would suggest that it may require a much longer treatment course to meaningfully effect inflammation in the airways.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No